CLINICAL TRIAL: NCT04402931
Title: Randomized Trial of Transcatheter Valve-in-Valve Intervention vs Redo Surgery for the Treatment of Structural Mitral Bioprosthetic Dysfunction
Brief Title: Randomized Trial of Transcatheter Valve-in-Valve vs Redo Surgery for Bioprosthetic Mitral Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Dante Pazzanese de Cardiologia (Other)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Principal Investigator, DIMYTRI ALEXANDRE DE ALVIM SIQUEIRA, Chief, Interventions in Acquired Valvular Heart Disease, Instituto Dante Pazzanese de Cardiologia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4993/2019
Record Dates: First submitted 2020-05-09; First posted 2020-05-27 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Mitral Prosthetic Valve Stenosis and Regurgitation
Keywords: Mitral Prosthetic valve dysfunction
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transcatheter Valve-in-Valve Intervention (Other): Transcatheter Valve-in-Valve Intervention
  Interventions: Procedure: Transcatheter Valve-in-Valve Intervention
- Redo Surgery (Other): Surgical Mitral valve replacement
  Interventions: Procedure: Redo Mitral valve surgery

INTERVENTIONS:
Procedure: Transcatheter Valve-in-Valve Intervention — Transcatheter mitral valve-in-valve implantation with SAPIEN 3
  Arms: Transcatheter Valve-in-Valve Intervention
Procedure: Redo Mitral valve surgery — Transcatheter Valve-in-Valve Intervention
  Arms: Redo Surgery

SUMMARY:
Transcatheter valve-in-valve implantation has emerged as a valid alternative to redo surgery for patients with surgical bioprosthetic dysfunction. Nowadays, transcatheter, transeptal mitral valve-in-valve replacement (TsMViV) has been adopted in many centers worldwide. Some studies report low rates of periprocedural morbidity and mortality and favorable hemodynamic parameters of valve performance. However, medium and long-term data on TsMViV as compared to redo surgical mitral valve replacement (rSMVR) is not yet established. Studies of cost-effectiveness and cost-utility comparing both strategies were also not reported. In particular, late prosthesis durability and hemodynamic performance after TsMViV are largely unknown and need to be elucidated before widely indicated, especially among younger and low-risk surgical candidates with failed mitral bioprostheses.

DETAILED DESCRIPTION:
Prospective, randomized, controlled trial of transeptal, transcatheter mitral valve-in-valve versus redo surgical mitral valve replacement.

After multidisciplinary, heart team discussion, patients meeting inclusion criteria will be randomized 1:1 to receive either transcatheter, transeptal mitral valve-in-valve replacement (TsMViV) with the SAPIEN 3 transcatheter heart valve (THV) or redo, mitral valve replacement with 3 commercially available surgical bioprosthetic valves. A sub-randomization in the surgical group will define which bioprosthetic valve will be used. Patients will be seen for follow-up visits at discharge, 30 days, 6 months and annually through 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years;
* Symptoms of heart failure NYHA class>ll;
* Severe mitral bioprosthetic dysfunction (stenosis, regurgitation, mixed) defined by echocardiography;
* Heart team (including cardiac surgeon) agree on eligibility including assessment that transeptal, transcatheter mitral valve replacement (TsMVR) and redo surgical mitral valve replacement (rSMVR) are appropriate;
* The study patient or the study patient's legal representative informed of the nature of the study, agreed to its provisions and provided written informed consent as approved by the Institutional Review Board (IRB) center;
* The study patient agreed to comply with all required post- procedure follow-up visits including annual visits through 10 years and analysis close date visits, which was conducted as a phone follow-up;
* Heart team agreed (a priori) on treatment strategy for concomitant coronary disease (if present);
* Patient agreed to undergo redo surgical mitral valve replacement (rSMVR) if randomized to control treatment.

Exclusion Criteria:

* Heart Team assessment of inoperability (including examining cardiac surgeon);
* Hostile chest;
* Evidence of an acute myocardial infarction < 1 month (30 days) before the intended treatment [defined as: Q wave Ml, or non-Q wave Ml with total creatine kinase (CK), creatine kinase MB isoform (CK-MB) and/or cardiac troponin elevations (WHO definition)];
* Concomitant severe valvular disease (aortic, tricuspid or pulmonic) requiring surgical intervention;
* Mitral mechanical prosthesis or mitral valve rings;
* Preexisting mechanical or bioprosthetic valve in other position with dysfunction;
* Complex coronary artery disease: unprotected left main coronary artery, Syntax score > 32 (in the absence of prior revascularization);
* Any therapeutic invasive cardiac procedure resulting in a permanent implant that is performed within 30 days of the index procedure (unless part of planned strategy for treatment of concomitant coronary artery disease). Implantation of a permanent pacemaker is not an exclusion criteria;
* Patients with planned concomitant surgical or transcatheter ablation for atrial fibrillation;
* Leukopenia (WBC < 3000 cell/mL), acute anemia (Hgb< 9 g/dL), thrombocytopenia (Pht< 50,000 cell/mL);
* Hypertrophic cardiomyopathy with or without obstruction (HOCM);
* Severe ventricular dysfunction with left-ventricular ejection fraction (LVEF) < 20%;
* Echocardiographic evidence of intracardiac mass, thrombus or vegetation;
* Active upper gastrointestinal (GI) bleeding within 3 months (90 days) prior to procedure;
* A known contraindication or hypersensitivity to all anticoagulation regimens, or inability to be anticoagulated for the study procedure;
* Clinically (by neurologist) or neuroimaging confirmed stroke or transient ischemic attack (TIA) within 3 months (90 days) of the procedure;
* Renal insufficiency (creatinine > 3.0 mg/dL) and/or renal replacement therapy at the time of screening;
* Estimated life expectancy < 24 months (730 days) due to carcinomas, chronic liver disease, chronic renal disease or chronic end stage pulmonary disease;
* Currently participating in an investigational drug or another device study;
* Active bacterial endocarditis within 6 months (180 days) of procedure;
* Patient refuses redo mitral valve replacement surgery.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Rate of Major cardiovascular and Cerebrovascular events | 12 months
  All-cause death; Cardiovascular death; Stroke

SECONDARY OUTCOMES:
Rate of Procedure-related complications | 30 days
  Major vascular complications;
  * Bleeding and transfusions;
  * Atrial fibrillation;
  * Acute renal failure;
  * Left-ventricular outflow obstruction;
  * Reoperation
Rate of Rehospitalization | 12 months
  Rehospitalization at 12 months
Rate of Prosthetic Thrombosis | 3 and 12 months
  Prosthetic thrombosis at 3- and 12 months (as assessed by transesophageal echocardiography and multi-slice tomography).
Rate of Structural Valve dysfunction (as assessed by transthoracic echocardiography) | 10 years
  Structural valve dysfunction assessed annually, up to 10-year follow-up.
Rate of Bioprosthetic Valve Failure (as assessed by clinical outcomes and echocardiographic evaluations) | 10 years
  Bioprosthetic valve failure assessed annually, up to 10-year follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Dimytri A Siqueira, MD, PhD, Principal Investigator — Instituto Dante Pazzanese de Cardiologia
Locations (7):
- Brazil (7):
  - Hospital de Messejana Dr. Carlos Alberto Studart Gomes, Fortaleza, Ceará
  - Hospital Ana Nery, Salvador, Estado de Bahia
  - Instituto Nacional de Cardiologia, Rio de Janeiro, Rio de Janeiro
  - Instituto de Cardiologia de Santa Catarina, São José, Santa Catarina
  - Instituto Dante Pazzanese de Cardiologia, São Paulo, São Paulo
  - UNIFESP, São Paulo, São Paulo
  - Instituto do Coração (INCOR), São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No